CLINICAL TRIAL: NCT00336674
Title: A Randomised, Double-blind, Placebo-controlled Trial of Intranasal Insulin (440 IU) in Children and Young Adults at Risk of Type 1 Diabetes: Intranasal Insulin Trial II
Brief Title: Trial of Intranasal Insulin in Children and Young Adults at Risk of Type 1 Diabetes
Acronym: INITII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INIT II
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DV001 (Active Comparator): Recombinant human intranasal insulin formulation in a buffered solution of benzalkonium chloride and glycerol presented in multi-dose nasal spray devices with actuators (Pfeiffer) designed to deliver 100ul spray doses to nasal mucosa. The product is formulated at a dose strength of 1100 IU / mL (40mg/mL) manufacturing formulation. The product will be self administered by eligible participants as two 100 microlitre spray doses per nostril. Treatment will be administered daily for 7 consecutive days then on one day each week for 12 months. Participants will be followed until they develop diabetes or until 5 years after the last participant has been randomised (maximum period of follow up is expected to be 10 years.
  Interventions: Biological: Intranasal insulin
- Placebo (Placebo Comparator): Placebo insulin carrier solution of benzalkonium chloride and glycerol presented in multi-dose nasal spray devices with actuators (Pfeiffer) designed to deliver 100ul spray doses to nasal mucosa. The product will be self administered by participants as two 100 microlitre spray doses per nostril. Treatment will be administered daily for 7 consecutive days then on one day each week for 12 months. Participants will be followed until they develop diabetes or until 5 years after the last participant has been randomised (maximum period of follow up is expected to be 10 years.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Intranasal insulin — 440IU Insulin
  Arms: DV001
Other: Placebo — Placebo insulin carrier solution containing benzalkonium chloride and glycerol
  Arms: Placebo

SUMMARY:
In people with type 1 diabetes the beta cells of the pancreas no longer make insulin because the body's immune system has attacked and destroyed the beta cells. It is thought that exposure of the mucous membranes to insulin may cause act like a vaccine effect whereby protective immune cells are stimulated and these then counteract the "bad" immune cells that damage the beta cells. This study aims to determine if intranasal insulin can protect beta cells and stop progression to diabetes in individuals who are at risk.

DETAILED DESCRIPTION:
Autoimmune diseases are the outcome of dysregulated immune responses to self-antigens. Type 1 diabetes (T1D), previously known as insulin-dependent or juvenile diabetes, is an autoimmune disease in which the body's immune system reacts against and destroys the insulin-producing β cells in the islets of the pancreas. T1D classically affects children and young adults. Approximately 15% of people with diabetes have this form of the disease and no treatment is currently available to prevent it. Asymptomatic individuals in the pre-clinical stage of T1D can be identified by the presence of circulating antibodies to the islet autoantigens (pro)insulin, glutamic acid decarboxylase (GAD) and tyrosine phosphatase-like insulinoma antigen 2 (IA2). (Pro)insulin is the only autoantigen that is specific for β cells and several lines of evidence demonstrate that it plays a key role in driving autoimmune β-cell destruction.

The ability to use self-antigens as tools to induce protective immunity, free from the side effects of conventional non-specific immunosuppression, is the 'Holy Grail' of autoimmune disease therapy. Animal models provide proof-of-concept for such antigen-specific therapy. For example, in the non-obese diabetic (NOD) mouse, a model of spontaneous T1D, transgenic over-expression of proinsulin in antigen-presenting cells in the immune system during development or in transferred bone marrow stem cells completely prevented diabetes. On a more practical and translatable level, immune tolerance to an antigen can be achieved by administering antigen to the mucosal immune system. Thus, immune responses to antigen are suppressed by feeding antigen ('oral tolerance') or by administering antigen to the naso-respiratory mucosa .

ELIGIBILITY:
Inclusion Criteria:

1. First-degree or second-degree relative of a person with Type 1 diabetes (T1D) diagnosed before age 40.
2. Age 4-30 years if first-degree relative; age 4-20 years if second-degree relative.
3. Confirmed serum antibodies to two or more islet antigens.
4. Normal oral glucose tolerance test (OGTT).
5. First phase insulin response (FPIR) at or above threshold - Primary Stratum - greater than or equal to 10th percentile for siblings, offspring and second-degree relatives of person with T1D (greater than or equal to 100uU/ml if aged 8 or more years OR greater than or equal to 60 uU/ml if aged less than 8) and greater than or equal to the 1st percentile for parents of someone with T1D (greater than ore equal to 60uU/ml). Secondary Stratum: Greater than or equal 1st percentile, less than 10th percentile for siblings, offspring and second-degree relatives of someone with T1D (greater than or equal to 50uU/ml less than 100 uU/ml if aged greater than or equal to 8 years or greater than or equal to 20 uU/ml less than 60uU/ml if aged less than 8 years)
6. Provision of written consent. -

Exclusion Criteria:

1. History of treatment with insulin or oral hypoglycemic agents
2. Known diabetes by ADA/WHO criteria
3. Pregnant or lactating or of child-bearing potential not using an adequate method of contraception
4. Concomitant disease or treatment which may interfere with assessment or cause immunosuppression, as judged by the investigators.
5. Uncorrected vitamin D deficiency
6. Known alcohol or drug abuse, psychiatric or other condition that could be associated with poor compliance.
7. Known liver disease, or persisting elevation of plasma Aspartate transaminase (AST) or Alanine transaminase (ALT) levels.
8. Impaired renal function
9. Any defect or pathology of nasal passage which would preclude application of the intranasal spray.

   -

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2006-12; Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Diabetes AT 5 years according to American Diabetes Association / World Health Organization (ADA/WHO) criteria. | 1 year of treatment 9 years follow up
  Defined as the presence of 2 or more of the following diagnostic criteria including diabetic fasting blood glucose level, diabetic 2 hour postprandial blood glucose level, diabetic HbA1c and symptoms

SECONDARY OUTCOMES:
B cell function | 1 year of treatment 9 years follow up
  Measured as glucose and insulin responses in Oral glucose tolerance test (OGTT) 6 monthly
Insulin Action | 1 year of treatment 9 years follow up
  Insulin resistance measured by Homeostasis of model assessment - resistance (HOMA-R) 6 monthly
Immune function | 1 year of treatment 9 years follow up
  Measured by levels of circulating antibodies to insulin, Glutamic acid decarboxylase (GAD) and Tyrosine phosphatase - like insulinoma antigen (IA-2) and T cell responses to proinsulin, denatured insulin, GAD and tetanus at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Leonard C Harrison, MBBS MD DSc, Principal Investigator — Melbourne Health
Locations (6):
- Australia (5):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Mater Children's Hospital, Brisbane, Queensland
  - Womens and Childrens Hospital, North Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Princess Margaret Hospital, Subiaco, Western Australia
- University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobsen LM, Schatz DA. Insulin immunotherapy for pretype 1 diabetes. Curr Opin Endocrinol Diabetes Obes. 2021 Aug 1;28(4):390-396. doi: 10.1097/MED.0000000000000648. PMID 34091488